CLINICAL TRIAL: NCT06725927
Title: Vaccination Against Influenza Pre-discharge in Patients Hospitalized Due to Heart Failure
Brief Title: Vaccination Against Influenza Pre-discharge in Heart Failure
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Michał Tkaczyszyn, MD, Dr, Wroclaw Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KB 659/2024
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure
Keywords: heart failure; influenza; vaccination
MeSH Terms: conditions — Heart Failure; Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Influenza vaccination (Experimental): Vaccination pre-discharge in patients stabilized after heart failure exacerbation
  Interventions: Biological: Influenza vaccination
- Standard of care (No Intervention)

INTERVENTIONS:
Biological: Influenza vaccination — Influenza vaccination pre-discharge in patients hospitalized due to heart failure exacerbation
  Arms: Influenza vaccination

SUMMARY:
In patients with heart failure (HF), influenza vaccination should be considered to prevent HF hospitalizations. However, vaccination rates among patients with HF are low, in part because of subjective but common concerns about whether patients with such severe disease should be vaccinated. In this randomized, open-label study, we will investigate whether influenza vaccination before discharge in patients stabilized after cardiac decompensation is safe and improves outcomes over a 6-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* informed consent to participate in the study
* hospitalization (unplanned) due to exacerbation (decompensation) of heart failure
* planned discharge within the next 48 hours due to completion of hospital treatment
* no current (2024/25 season) influenza vaccination.

Exclusion Criteria:

* severe post-vaccination reaction during influenza vaccination in any previous influenza season
* hypersensitivity to any of the components of the vaccine planned to be administered
* discharge to another hospital for continued treatment or discharge to a nursing home
* antibiotic therapy among the drugs recommended for taking after hospitalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Primary composite endpoint - cardiovascular death, heart failure hospitalization or infection | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jan Biegus, Professor, Study Chair — Wroclaw Medical University
Locations (1):
- Jan Mikulicz Radecki University Hospital in Wroclaw, Wroclaw, Lower Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No